CLINICAL TRIAL: NCT03576950
Title: Uterine Rupture in Pregnancy: the URIDA (Uterine Rupture International Data Acquisition) Study
Brief Title: Uterine Rupture International Data Acquisition
Acronym: URIDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, Università degli Studi dell'Insubria
Other Study IDs: URIDA
Record Dates: First submitted 2018-06-21; First posted 2018-07-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Uterine Rupture Gravid
Keywords: Uterine rupture; Cesarean section; Labour; Myomectomy; Delivery
MeSH Terms: conditions — Uterine Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uterine rupture: Women with uterine rupture occurred during pregnancy.

SUMMARY:
Uterine rupture represents an uncommon event: it is is a life-threatening obstetric complication with high maternal and perinatal morbidity and mortality. Indeed, uterine rupture may cause catastrophic maternal and fetal complications (uterine hemorrhage, hysterectomy with consequent fertility loss, maternal and fetal death or cerebral palsy) which are hardly acceptable within the context of a natural event such as birth.

Uterine rupture can occur during pregnancy, early in labor or following a prolonged labor, most frequently near or at term and, rarely, during early to mid-pregnancy. Its prevalence ranges between 0.006% for women without previous cesarean section (CS) in the western countries, to 25% for women with obstructed labor in African countries.

Pregnancy after myomectomy or CS, vaginal delivery after cesarean sections (VBACs) and vaginal delivery after myomectomy are potentially "at risk" of uterine rupture.

Despite uterine rupture is widely considered a life-threatening condition, so far most of published data refer to case reports or very small case series. In this scenario, the "Uterine Rupture International Data Acquisition" study group would like to collect a large number of events, in order to identify the potential risk factors among different populations through a multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women with uterine rupture occurred during pregnancy.

Exclusion Criteria:

* None.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Women with uterine rupture occurred during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Uterine rupture | A retrospective analysis of 10 years.
  Women with uterine rupture occurred during pregnancy.

SECONDARY OUTCOMES:
Gestational age at uterine rupture | A retrospective analysis of 10 years.
  Gestational age, calculated as weeks and days, in which uterine rupture occurred.
Parity | A retrospective analysis of 10 years.
  The number of previous delivery.
Body Mass Index | A retrospective analysis of 10 years.
  The Body Mass Index of each patient in which uterine rupture occurred.
Presence of myomas | A retrospective analysis of 10 years.
  The occurrence of myomas in each patient in which uterine rupture occurred.
Hysterectomy | A retrospective analysis of 10 years.
  The number of cases in which it was necessary to perform hysterectomy after uterine rupture.
Hospital stay | A retrospective analysis of 10 years.
  The hospital stay from the admission to the discharge, expressed in days.
Neonatal complications | A retrospective analysis of 10 years.
  The occurrence of neonatal complications, included neonatal deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tinelli, M.D., Study Director — U.O. Ginecologia e Ostetricia, Ospedale Vito Fazzi, 73100 Lecce, Italy

IPD SHARING:
Plan to Share IPD: Undecided